CLINICAL TRIAL: NCT05408104
Title: Postoperative Tolvaptan Use in Left Ventricular Assist Device Implantation Patients
Acronym: TOLVAD
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB19-0111
Record Dates: First submitted 2022-05-24; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure; Heart Assist Device; Hyponatremic
Keywords: Tolvaptan
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tolvaptan (TLV): LVAD recipients with post-operative hyponatremia (Na < 135 mEq/L). Eligible patients took tolvaptan 15 mg daily as part of a routine care treatment plan.
  Interventions: Drug: tolvaptan
- no tolvapton (no-TLV): LVAD recipients with post-operative hyponatremia (Na < 135 mEq/L). Eligible patients did not take tolvaptan as part of routine care.

INTERVENTIONS:
Drug: tolvaptan — LVAD recipients with post-operative hyponatremia (Na < 135 mEq/L). Subjects took tolvaptan 15 mg daily as part of their standard care.
  Groups: tolvaptan (TLV)

SUMMARY:
This research study will compare two standard of care approaches for managing low sodium levels in heart failure patients with Left Ventricular Assist Device (LVAD). The study will compare the outcomes of LVAD patients with low sodium levels who take Tolvaptan to those who do not take Tolvaptan. Tolvaptan is FDA approved for use in the study population and is commonly used to treat low sodium levels in heart failure and LVAD patients. It is not known if taking Tolvaptan or not taking Tolvaptan is better at improving outcomes in newly implanted LVAD patients with low sodium levels. By doing this study, the Principal Investigator (PI) hopes to learn which is better at improving outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with American College of Cardiology (ACC) and the American Heart Association (AHA) Stage D heart failure and plan to undergo LVAD implantation
* Age greater than or equal to 18 years old

Exclusion Criteria:

* No plan for LVAD implantation
* Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients at University of Chicago Medical Center (UCMC) being followed by the advanced heart failure group that are planned to undergo LVAD implantation.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Increase in Na level from the first post-operative day of hyponatremia, defined as Na < 135 mEq/L, to one-month follow-up. | one month
Change in renal function, measured by estimated glomerular filtration rate (eGFR), from first post-operative day to one-month follow-up. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Gene Kim, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States